CLINICAL TRIAL: NCT06323616
Title: The Effect of Anesthesia Depth Monitoring on Emergence Agitation and Delirium in Pediatrics
Brief Title: The Effect of Anesthesia Depth Monitoring on Emergence Delirium in Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Meltem Savran Karadeniz, Associate Professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2023/2343
Record Dates: First submitted 2024-03-15; First posted 2024-03-21 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2024-07

CONDITIONS: Anesthesia; Emergence Delirium; Anesthesia Awareness; Behavior Child Problems; Postoperative Delirium; Postoperative Complications
MeSH Terms: conditions — Emergence Delirium; Intraoperative Awareness; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Randomized, Single-Blind, Prospective, Interventional
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): Sevoflurane anesthesia will be applied with an endtidal agent consumption of 0.8 MACage, with 2 standard deviations for MACage:1 to the control group, as we apply in routine anesthesia practice. (During the surgery, the parameters showing the depth of anesthesia will be placed away from the anesthesiologist and covered to ensure blindness. At the end of the surgery, the data will be received via USB.)
- Study Group (Experimental): Sevoflurane anesthesia will be applied to the study group by adjusting the MAC to keep the PSI median value between 25-50 (if PSI<25, MAC will be reduced by 0.1, if PSI>50, MAC will be increased by 0.1).
  Interventions: Procedure: MAC adjustment to PSI between 25 and 50

INTERVENTIONS:
Procedure: MAC adjustment to PSI between 25 and 50 — According to SedLine monitoring, the depth of anesthesia will be adjusted by changing the amount of sevoflurane so that the PSI median value is between 25 and 50.
  Arms: Study Group

SUMMARY:
Some changes in the patient's cognitive state are observed during the recovery period from general anesthesia. This period of behavioral dysregulation has been called emergence agitation (EA) and emergence delirium (ED). ED and EA occur in the early postoperative period (often within the first 30 minutes). The incidence of ED ranges from 10% to 80% in children and is described as a distressing clinical condition by 42% of pediatric anesthesiologists. Self-harm by the child increases the risk of delayed discharge and may increase the cost of medical care.

Sevoflurane is a widely used agent for the induction and maintenance of anesthesia, but its use is associated with the occurrence of ED in the pediatric population. Clinical findings are characterized by hallucinations, struggling, restlessness, crying, and disorientation.

In the literature, the Pediatric Anesthesia Rescue Delirium (PAED) Scale Score is used in the diagnosis of ED and EA. This score consists of 5 criteria (maximum score 20) scored using 0-4 point scales. These criteria; The child needs to make eye contact with the caregiver, the child's movements are purposeful, the child is aware of the environment, the child is restless/angry, the child cannot be consoled. While the sensitivity of ≥10 points for the diagnosis of ED is 64% and the specificity is 86%, the sensitivity of >12 points for the diagnosis of ED is 100% and the specificity is 94.5%.

Monitoring intraoperative depth of anesthesia in the adult population has been recommended by the American Society of Anesthesiologists (ASA) due to its potential benefits such as faster recovery time and lower drug dosage, as well as prevention of adverse effects such as the incidence of hypotension. The use of anesthesia depth monitors used so far for children is controversial because brain development in children has not yet been completed and the calculation algorithms of these indices are based on adult EEG characteristics.

There are very few studies in the literature on the relationship between anesthesia depth monitoring and EA/ED in children, and further studies are needed.

DETAILED DESCRIPTION:
During the compilation period after general anesthesia, cognitive status changes called emergence agitation and emergence delirium, clinically characterized by hallucinations, struggling, restlessness, crying, and disorientation, are observed. ED and EA often occur in the early postoperative period (especially in the first 30 minutes).

Sevoflurane is a widely used agent for the induction and maintenance of anesthesia, but its use is associated with the occurrence of ED/EA in the pediatric population. In our study, we aimed to determine the effect of sevoflurane anesthesia on the incidence of ED/EA under anesthesia depth monitoring.

Patients who give informed consent will be divided into 2 groups and randomized using the opaque sealed envelope method.

Children participating in the study will be evaluated with mYPAS, an anxiety assessment scale, in the preoperative period. Studies have found that children with high levels of anxiety have a higher frequency of developing maladaptive behavioral changes, pain, and ED after surgery.

On the day of surgery, patients will be taken to the operating room after premedication with 0.5 mg/kg po midazolam. Following routine noninvasive blood pressure, saturation and ECG monitoring; PEEG monitoring will be carried out with the help of pediatric sensors. Anesthesia guided by PEEG (processed electroencephalography) contributes to optimal targeting of the depth of anesthesia. The rationale for PEEG is to provide a simplified method for monitoring the depth of anesthesia through rapid interpretation of the frontal electroencephalogram (EEG). Thus, 4-channel raw EEG (L1, R1, L2 and R2 - equivalent to Fp1, F7, Fp2 and F8 according to the standard EEG monitoring system), electrode impedance, patient condition index (PSI), left and right spectral edge frequency (SEF95) and burst suppression ratio (SR) can be achieved. PSI; It is a dimensionless depth of anesthesia index that combines "weighted quantitative EEG parameters reflecting multiple dimensions of brain electrical activity." The correct depth of anesthesia is determined by the PSI value between 25 and 50.

Following inhaler induction with 8% sevoflurane, 0.5 mg/kg rocuronium and 2 mcg/kg fentanyl will be administered iv. Anesthesia maintenance of the patients will be provided with sevoflurane and 0.02-0.1mcg/kg/min remifentanil iv infusion.

To the control group; As we apply in routine anesthesia practice, sevoflurane anesthesia will be applied with Endtidal agent consumption of 0.8 MACage for MACage:1 with 2 standard deviations. During the surgery, parameters indicating the depth of anesthesia will be placed away from the anesthesiologist and closed to ensure blindness. At the end of the surgery, the data will be received via USB.

As for the working group; Sevoflurane anesthesia will be applied by adjusting the MAC so that the PSI median value remains between 25-50 (if PSI<25, MAC will be reduced by 0.1, if PSI>50, MAC will be increased by 0.1).

At the end of inhalation anesthesia, regional anesthesia (peripheral nerve/body block) will be applied to both groups for postoperative analgesia.

At the end of the operation, the PAED scores of all children 5, 15 and 30 minutes after extubation will be evaluated and recorded by PACU (post-anesthesia care unit) nurses who are blind to the study groups.

Ped-PADSS score, defined as the discharge score, will be checked at 30, 45 and 60 minutes in the compilation room. This score consists of 5 criteria which are vital signs, activity level, nausea-vomiting, presence of pain (<6 years OPS, >6 years VAS) and surgical bleeding. It is evaluated between 0 and 10 points, 9 points and above are safe for discharge from the compilation room.

In the post-hospital discharge period, the PHBQ scale will be administered to patients via an online survey on days 3, 14 and 28. This scale is a post-discharge behavior scale developed for children, consisting of six subscales (general anxiety, separation anxiety, sleep, eating, aggression, apathy) and 27 questions. Values between 27-135 points will be recorded and evaluated in terms of whether late-term behavioral changes occur.

There is little data in the literature on the relationship between anesthesia depth monitoring and ED during recovery in children, and further studies are needed. In our study, we think that the frequency of ED will be less in the study group than in the control group.

ELIGIBILITY:
Inclusion Criteria:

* 2 to 8 years old
* Surgery time > 1 hour
* Urology, Plastic Surgery and Pediatric Surgery patients

Exclusion Criteria:

* Patients with neuromotor development abnormalities
* Patients with a history of epilepsy/antiepileptic treatment
* Patients receiving intraoperative ketamine administration
* Patients requiring postoperative ICU admission
* Surgeries performed under emergency conditions
* Patients without parental consent

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2024-02-22 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
ED/EA incidence | postoperative 5th, 15th and 30th minutes
  The Pediatric Anesthesia Recovery Delirium (PAED) Scale Score will be used. This score consists of 5 criteria (maximum score 20) scored using 0-4 point scales. These criteria; The child must make eye contact with the caregiver, the child's movements are purposeful, the child is aware of the surroundings, the child is restless/irritable, and the child cannot be consoled. A score of ≥10 will be considered EA, and a score of >12 will be considered ED.

SECONDARY OUTCOMES:
mYPAS | immediately before induction of anesthesia
  The mYPAS is an observational measure of children's preoperative anxiety consisting of 27 items divided into 5 categories: Activity, Vocalizations, Emotional Expressivity, State of Arousal and Use of Parent. Ratings produce 4 mYPAS scores (1 for each time point). Each score is calculated by dividing each item rating by the highest possible rating (i.e., 6 for the 'vocalizations' item and 4 for all other items), adding all of the produced values, dividing by 5, and multiplying by 100. This calculation produces a score ranging from 23.33 to 100 with higher values indicating higher anxiety.
PSI <25 episode duration | intraoperative
  The duration of PSI <25 throughout the surgery will be calculated by looking at the trend table at the end of the surgery on the sedLine monitor.
PSI >50 episode duration | intraoperative
  The duration of PSI >50 throughout the surgery will be calculated by looking at the trend table at the end of the surgery on the sedLine monitor.
PSI <25 number of episodes | intraoperative
  If PSI <25 is observed within 15 minutes, it will be noted as an episode. More than one PSI <25 cases observed within the same 15 minutes will be included in the same episode and counted as a single episode.
PSI >50 number of episodes | intraoperative
  If PSI >50 is observed within 15 minutes, it will be noted as an episode. More than one PSI >50 cases observed within the same 15 minutes will be included in the same episode and counted as a single episode.
Suppresyon ratio | intraoperatively every 15 minutes
  The SR (Supration Ratio) parameter, which shows the depth of suppressed anesthesia on the SedLine monitor, will be recorded
SEF95R | intraoperatively every 15 minutes
  The right spectral edge frequency (SEF95R) value on the SedLine monitor will be recorded every 15 minutes
SEF95L | intraoperatively every 15 minutes
  The left spectral edge frequency (SEF95L) value on the SedLine monitor will be recorded every 15 minutes
Mean blood pressure | intraoperatively every 15 minutes
  non invasive blood pressure measurement
Heart rate | intraoperatively every 15 minutes
  ECG monitoring
SpO2 | intraoperatively every 15 minutes
  pulse oximeter
Total amount of sevoflurane used | at the end of surgery
  At the end of the surgery, the number of milliliters will be recorded by looking at the trend parameters on the anesthesia device.
Total amount of remifentanil used | at the end of surgery
  At the end of the surgery, the total number of micrograms from the infusion pump will be recorded.
MAC | intraoperatively every 15 minutes
  The MACage value on the anesthesia device will be recorded every 15 minutes throughout the surgery.
Waking up time | at the end of surgery
  The time between the end of sevoflurane anesthesia and eye opening will be recorded with a stopwatch.
Pupil size | intraoperatively every 15 minutes
  3 points will be recorded as mydriasis, 1 point as miosis, and values between will be recorded as 2 points every 15 minutes.
Anesthesia duration | perioperative
  The time between induction and awakening will be recorded using a stopwatch.
Surgery duration | perioperative
  The time between the start and end of surgery will be recorded with the help of a stopwatch.
PHBQ | postoperative 3rd, 14th and 28th day
  In the period after discharge from the hospital, PHBQ (The Post Hospitalization Behavior Questionnaire) will be sent to patients via an online survey on days 3, 14 and 28. This questionnaire is a post-discharge behavior form developed for children consisting of six subscales (general anxiety, separation anxiety, sleep, eating, aggression, apathy) and 27 questions. Values between 27-135 points will be evaluated according to the record in terms of whether the change in the transition period has developed or not.
Ped-PADS | postoperative 30th, 45th and 60th minutes
  The Ped-PADSS score, defined as the discharge score, will be checked by the recovery nurses at the 30th, 45th and 60th minutes. This score consists of 5 criteria (vital signs, activity level, nausea and vomiting, presence of pain (<6 years OPS, >6 years VAS) and surgical bleeding. It is evaluated between 0 and 10 points. A score of 9 points and above is safe for discharge from the recovery room. .
Time of discharge from hospital | 14 days after operation
  It will be learned and recorded by calling 14 days after the operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Murray HW, Soave R. Appendicitis with perforation: a reminder to internists. South Med J. 1980 Jun;73(6):730-1. doi: 10.1097/00007611-198006000-00013. PMID 7394591
- [Background] Ricci Z, Robino C, Rufini P, Cumbo S, Cavallini S, Gobbi L, Brocchi A, Serio P, Romagnoli S. Monitoring anesthesia depth with patient state index during pediatric surgery. Paediatr Anaesth. 2023 Oct;33(10):855-861. doi: 10.1111/pan.14711. Epub 2023 Jun 19. PMID 37334678
- [Background] Kain ZN, Caldwell-Andrews AA, Maranets I, McClain B, Gaal D, Mayes LC, Feng R, Zhang H. Preoperative anxiety and emergence delirium and postoperative maladaptive behaviors. Anesth Analg. 2004 Dec;99(6):1648-1654. doi: 10.1213/01.ANE.0000136471.36680.97. PMID 15562048